CLINICAL TRIAL: NCT04909749
Title: CDDOM Oneome Rightmed Depression Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Collaborators: OneOme, LLC (Industry)
Responsible Party: Principal Investigator, Lawrence Mandarino, Professor, Division Chief, CDDOM Director, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1901270218
Record Dates: First submitted 2020-07-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Approximately 100,000 patients are clinically managed by El Rio providers each year. A PHQ-2 is routinely completed by all visiting patients at El Rio health to screen for depression. Patients who screen positive on the PHQ-2 subsequently take the PHQ-9, a similar but more sensitive and specific depression assessment tool. For our study, a total of 350 patients will be recruited and randomized to PGx-guided antidepressant therapy (n= 175) or treatment as usual (n =175). Patients who are currently clinically managed for depression will be eligible for participation as well. Patients who are pregnant, have a history of major depressive disorder, or a concurrent diagnosis of other psychiatric issues will be excluded. Patients who will not be treated with antidepressants will be excluded
Who Masked: Participant, Investigator
Masking Description: Primary study Investigator(s) and analyzers of samples with be masked. Only one co-I responsible for group randomization will be unmasked to study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGx-guided antidepressant therapy (Experimental): These individuals will be prescribed medication guided by the Oneome RightMed Test.
  Interventions: Genetic: Oneome RightMEd Pharmacogenomic testing Kit
- Treat as usual based on Clinical Physician Recommendation (No Intervention): These individuals will receiving medication as usual based on the clinics internal guidelines and physician recommendations.

INTERVENTIONS:
Genetic: Oneome RightMEd Pharmacogenomic testing Kit — The RightMed test is an end-to-end solution which includes sample collection, pharmacogenomic (PGx) testing services, data analysis, and clinical interpretation that helps physicians select treatments based on evidence-driven predictions of patient drug response and tolerance. Genetic components of an individual's drug response are well established and often included on Food and Drug Administration (FDA) medication labels. The OneOme RightMed test has incorporated existing evidence to classify the risk and likelihood of an antidepressant working for different patients. Patient results for each medication can fall into one of three categories: 1.) Green - use as directed; 2.) Yellow - use with caution; and 3.) Red - adjust dose or choose alternative mediation and can be used proactively or reactively
  Arms: PGx-guided antidepressant therapy

SUMMARY:
In this study, we hypothesize PGx guided testing can improve outcomes related to treatment of moderate and severe depression among El Rio Community Health patients. We anticipate patients randomized to the OneOme RightMed® PGx test will demonstrate a greater improvement of depressive symptoms and will have a higher proportion of subjects reporting response and remission than those receiving standard care.

Our purpose is to determine the effectiveness and feasibility of implementing a pharmacogenomic (PGx) approach to prescribing antidepressant medication in an underserved, community health center patient population.

DETAILED DESCRIPTION:
In this study, we hypothesize PGx guided testing can improve outcomes related to treatment of moderate and severe depression among El Rio Community Health patients. We anticipate patients randomized to the OneOme RightMed® PGx test will demonstrate a greater improvement of depressive symptoms and will have a higher proportion of subjects reporting response and remission than those receiving standard care.

Our purpose is to determine the effectiveness and feasibility of implementing a pharmacogenomic (PGx) approach to prescribing antidepressant medication in an underserved, community health center patient population.

Primary Outcomes:

1. Changes in patient depressive ratings will be the primary endpoint in this study. The primary outcome will be measured using the validated Patient Health Questionnaire (PHQ-9) depression rating scale, administered verbally to participants.

   Depression response and remission rates (proportion of subjects achieving or not achieving), in the control and intervention arm will be directly compared at baseline, 2, 4, 8, and 12 weeks.
2. Patient progression from primary care to El Rio behavioral health (BH) specialty care will also be monitored in this study. We will directly compare the proportion of subjects in the control and intervention arm requiring BH consultation at any point in the study.

Secondary Outcomes:

1. Medication changes - Number of antidepressant medication changes and/or dose adjustments per subject from baseline to study endpoint.
2. Medication congruence - Alignment of physicians to RightMed test recommendations in control and intervention arm (guided vs unguided) and time to achieve optimal medication selection (green bin).

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* PHQ-9 score ≥ 10
* Suffer from Major Depressive Disorder meeting DSM-V criteria and meet at least one of the following:

  * Either new to antidepressant treatment or currently taking medication for less than 6 weeks.
  * Inadequate efficacy after at least 6 weeks of antidepressant treatment
  * Have discontinued antidepressant treatment due to adverse events or intolerability within the last 6 weeks
* Must be able to understand requirements of the study and provide written informed consent (English or Spanish)

Exclusion Criteria:

* Any patient for whom providing a buccal swab sample would be contraindicated or not possible.
* Patients taking antidepressants for > 6 months consecutively prior to baseline unless determined to be inadequate efficacy and PCP looking to change medication.
* Subjects diagnosed as not having or depression.
* Patients with history of prior PGx testing
* Inability to provide informed consent
* Current diagnosis of bipolar disorder type I or II, psychosis, schizophrenia and/or schizoaffective disorder
* Inability to attend scheduled study visits
* Patients who are known to be pregnant or lactating
* Patients that are diagnosed with severe depression

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
determine the effectiveness and feasibility of implementing a pharmacogenomic (PGx) approach to prescribing antidepressant medication | 2 years
  Our purpose is to determine the effectiveness and feasibility of implementing a pharmacogenomic (PGx) approach to prescribing antidepressant medication in an underserved, community health center patient population
  1.) Changes in patient depressive ratings will be the primary endpoint in this study. The primary outcome will be measured using the validated Patient Health Questionnaire (PHQ-9) depression rating scale, administered verbally to participants.

IPD SHARING:
Plan to Share IPD: No
Individual results (IPD) will not be shared.